CLINICAL TRIAL: NCT02576431
Title: A Study to Learn How Well the Drug Larotrectinib Works in Adults With Different Solid Cancers With a Change in the Genes Called NTRK Fusion
Brief Title: A Study to Test the Effect of the Drug Larotrectinib in Adults and Children With NTRK-fusion Positive Solid Tumors
Acronym: NAVIGATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20289; LOXO-TRK-15002 (Other: Loxo Oncology, Inc); 2022-502667-38-00 (Other: CTIS (EU)); 2015-003582-28 (EudraCT Number)
Expanded Access: NCT03025360 (Approved for marketing)
Record Dates: First submitted 2015-10-12; First posted 2015-10-15 (Estimated); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumors Harboring NTRK Fusion
Keywords: Non-small cell lung cancer; Thyroid cancer; Sarcoma; Colorectal cancer; Salivary gland cancer; Biliary cancer; Central nervous system (CNS) Tumor; Breast cancer; Melanoma; Neurotrophic tyrosine receptor kinase (NTRK); NTRK1; NTRK2; NTRK3; Fusion Positive; TRK fusion; TRKA; TRKB; TRKC; ETV6
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Thyroid Neoplasms; Sarcoma; Colorectal Neoplasms; Salivary Gland Neoplasms; Biliary Tract Neoplasms; Neoplasms; Breast Neoplasms; Melanoma | interventions — larotrectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Arm 1_NSCLC (Experimental): Patients with solid non-small cell lung cancer (NSCLC) harboring NTRK fusions (arm closed)
  Interventions: Drug: BAY2757556 (Larotrectinib, Vitrakvi)
- Arm 2_Thyroid (Experimental): Patients with solid thyroid tumors harboring NTRK fusions (arm closed)
  Interventions: Drug: BAY2757556 (Larotrectinib, Vitrakvi)
- Arm 3_Sarcoma (Experimental): Patients with soft-tissue sarcoma harboring NTRK fusions (arm closed)
  Interventions: Drug: BAY2757556 (Larotrectinib, Vitrakvi)
- Arm 4_Colorectal (Experimental): Patients with solid colorectal tumors harboring NTRK fusions (arm closed)
  Interventions: Drug: BAY2757556 (Larotrectinib, Vitrakvi)
- Arm 5_Salivary (Experimental): Patients with solid salivary tumors harboring NTRK fusions (arm closed)
  Interventions: Drug: BAY2757556 (Larotrectinib, Vitrakvi)
- Arm 6_Biliary (Experimental): Patients with solid biliary tumors harboring NTRK fusions (arm closed)
  Interventions: Drug: BAY2757556 (Larotrectinib, Vitrakvi)
- Arm 7_Primary CNS (Experimental): Patients with solid tumors in the primary central nervous system (CNS) harboring NTRK fusions (arm closed)
  Interventions: Drug: BAY2757556 (Larotrectinib, Vitrakvi)
- Arm 8_Other tumors (Experimental): Patients with e.g. kidney cancer, squamous cell cancer of head or neck or ovarian solid tumors harboring NTRK fusions (arm closed)
  Interventions: Drug: BAY2757556 (Larotrectinib, Vitrakvi)
- Arm 9_Solid tumors without confirmed NTRK fusion (Experimental): Patients eligible for arms 1 to 8, but with documented NTRK fusion from a laboratory where CLIA or equivalent certification cannot be confirmed by the sponsor at the time of consent (arm closed)
  Interventions: Drug: BAY2757556 (Larotrectinib, Vitrakvi)
- Arm 10_Prospective cohort (Experimental): Patients with melanoma, non secretory breast and colorectal cancer or other tumor types harboring NTRK fusions, except soft tissue sarcoma, salivary gland and thyroid cancer (arm closed)
  Interventions: Drug: BAY2757556 (Larotrectinib, Vitrakvi)
- Arm 11_Bone health cohort (Experimental): Patients with all tumor types harboring NTRK fusions, not eligible for the main prospective cohort, including patients with non-measurable disease
  Interventions: Drug: BAY2757556 (Larotrectinib, Vitrakvi)

INTERVENTIONS:
Drug: BAY2757556 (Larotrectinib, Vitrakvi) — Larotrectinib will be administered orally as capsule or liquid solution at a dose of 100 mg twice daily in continuing 28-days cycles.
  Other Names: LOXO-101

SUMMARY:
This research study is done to test how well different types of cancer respond to the drug called larotrectinib. The cancer must have a change in a particular gene (NTRK1, NTRK2 or NTRK3). Larotrectinib is a drug that blocks the actions of these NTRK genes in cancer cells and can therefore be used to treat cancer.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the efficacy of larotrectinib for the treatment of advanced solid tumors harboring a fusion of neurotrophic tyrosine receptor kinase (NTRK) of types 1-3 in children and adults.

Secondary objectives comprise the efficacy and safety of larotrectinib in different NTRK-tumor types.

ELIGIBILITY:
Inclusion Criteria:

* Locally-advanced or metastatic malignancy with an NTRK1, NTRK2, or NTRK3 gene fusion, identified through molecular assays as routinely performed at CLIA or other similarly-certified laboratories. Subjects who have an NTRK gene fusion identified in a lab where CLIA or equivalent certification cannot be confirmed by the Sponsor at the time of consent may have been enrolled in Cohort 9 as per protocol versions 1.0 - 8.0. From protocol version 9.0: CLIA or similar certification of the lab performing the fusion assay is required. However, patients may be included after discussion with the sponsor if the lab performing the fusion assay is not CLIA or similar certified.
* Subjects who have received prior standard therapy appropriate for their tumor type and stage of disease, or who have no satisfactory alternative treatments and in the opinion of the Investigator, would be unlikely to tolerate or derive clinically meaningful benefit from appropriate standard of care therapy.
* Subjects must have at least one measurable lesion as defined by RECIST v1.1 (Eisenhauer et al. 2009). Subjects with solid tumors without RECIST v1.1 measurable disease (e.g., evaluable disease only) had been eligible for enrollment to Cohort 8 as per protocol versions 1.0 - 8.0, regardless of tumor type. Subjects with primary CNS tumors should meet the following criteria:

  1. Have received prior treatment including radiation and/or chemotherapy, with radiation completed > 12 weeks prior to C1D1 of therapy, as recommended or appropriate for that CNS tumor type.
  2. Have ≥ 1 site of bi-dimensionally measurable disease (confirmed by magnetic resonance imaging [MRI] and evaluable by RANO criteria), with the size of at least one of the measurable lesions ≥ 1 cm in each dimension and noted on more than one imaging slice.
  3. Imaging study performed within 28 days before enrollment. If on steroid therapy, the dose must be stable for at least 7 days immediately before and during the imaging study.
  4. Must be neurologically stable based on stable neurologic exam for 7 days prior to enrollment.

     For subjects eligible for enrollment to bone health cohort, inclusion criterion 3 is modified as the following:
  5. Subjects must have at least one lesion at baseline (measurable or non-measurable as defined by RECIST v1.1 or RANO criteria, as appropriate to tumor type).
  6. Subjects with primary CNS tumors must be neurologically stable based on stable neurologic exam for 7 days prior to enrollment.
* At least 18 years of age
* Performance Status: Eastern Cooperative Oncology Group (ECOG) score ≤ 3. If enrolled with primary CNS tumor to be assessed by RANO, Karnofsky Performance Score (KPS) ≥ 50%.
* Tumor tissue before treatment (mandatory). If neither fresh tissue can be obtained nor archival tissue is available patients might be enrolled after consultation with the sponsor.
* Adequate organ function as defined by the following criteria:

  1. Serum AST and serum ALT < 2.5 x upper limit of normal (ULN), or AST and ALT < 5 x ULN if liver function abnormalities are due to underlying malignancy
  2. Total bilirubin < 2.5 x ULN, except in the setting of biliary obstruction. Subjects with a known history of Gilberts Disease and an isolated elevation of indirect bilirubin are eligible
  3. Serum creatinine < 2.0 x ULN OR an estimated glomerular filtration rate ≥ 30 mL/minute using the Cockcroft-Gault formula: (140- age) x body weight (kg) x 0.85 (if female)/serum creatinine (mg/dL) x 72 with either result acceptable for enrollment.
* Ability to comply (or for guardian to ensure compliance) with outpatient treatment, laboratory monitoring, and required clinic visits for the duration of study participation.
* Willingness of men and women of reproductive potential to use double effective birth control methods, defined as one used by the subject and another by his/her partner, for the duration of treatment and for 1 month following study completion.
* For subjects eligible for enrollment to bone health cohort only: life expectancy of at least 6 months, based on investigator assessment.

Exclusion Criteria:

* Investigational agent or anticancer therapy within 2 weeks prior to the planned start of larotrectinib or 5 half-lives, whichever is shorter, and without recovery of acute and/or clinically significant toxicities from that therapy.
* Prior progression while receiving approved or investigational tyrosine kinase inhibitors targeting TRK. Subjects who received less than 28 days of treatment and discontinued because of intolerance or toxicity are eligible.
* Symptomatic or unstable brain metastases. (Note: Subjects with asymptomatic brain metastases are eligible to participate in the study.) Subjects with primary CNS tumors are eligible.
* Uncontrolled concurrent malignancy that would limit assessment of efficacy of larotrectinib. Allowed conditions may include, but are not limited to in situ cancers of cervix, breast, or skin, superficial bladder cancer, limited-stage prostate cancer, and basal or squamous cancers of the skin.
* Active uncontrolled systemic bacterial, viral, or fungal infection CTCAE grade ≥ 2; unstable cardiovascular disease, or other systemic disease that would limit compliance with study procedures. Unstable cardiovascular disease is defined as:

  1. In adults, persistently uncontrolled hypertension defined as systolic blood pressure (BP) > 150 mmHg and/or diastolic BP > 100 mmHg despite antihypertensive therapy.
  2. Myocardial infarction within 3 months of screening.
  3. Stroke within 3 months of screening.
* Inability to discontinue treatment with a strong CYP3A4 inhibitor or inducer
* Currently recovering from AEs/ ADRs due to previous treatments (excluding alopecia). Inclusion is only advised once the AE/ADR resolves or recovers to baseline or at least to CTCAE grade 1.
* Known or suspected hypersensitivity against the active substance or any of the ingredients of the IMP.
* Known history of HIV infection. All patients must be screened for HIV up to 28 days prior to study drug start using a blood test for HIV according to local regulations.
* HBV or HCV infection. All patients must be screened for HBV and HCV up to 28 days prior to study drug start using the routine hepatitis virus laboratorial panel. Patients positive for HBsAg or HBcAb will be eligible if they are negative for HBVDNA. Patients positive for anti-HCV antibody will be eligible if they are negative for HCV-RNA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Best overall response of confirmed complete response (CR) or partial response (PR) as determined by an independent radiology review committee using RECIST v1.1 or RANO criteria, as appropriate to tumor type. | Up to 120 months

SECONDARY OUTCOMES:
Best overall response of confirmed CR or PR as determined by the treating Investigator using RECIST v1.1 or RANO criteria, as appropriate to tumor type | Up to 120 months
Duration of response (DOR): determined for subjects with best overall response of confirmed CR or PR by 1) an independent radiology review committee and 2) the treating Investigator | Up to 120 months
  Duration of response is the number of months from the start of confirmed complete response or partial response to disease progression or death. Complete response, partial response and disease progression are assessed by an independent radiology committee (IRC).
Clinical benefit rate (CBR): best overall response of confirmed CR, PR, or stable disease lasting 16 or more weeks following the initiation of Larotrectinib | Up to 120 months
Rate of subjects that have any tumor regression as a best response, measured as shrinkage of target lesions | Up to 120 months
PFS: Number of months from initiation of larotrectinib to the earlier of disease progression or death due to any cause | Up to 120 months
Overall Survival (OS): Number of months from the initiation of larotrectinib to the date of death due to any cause. | Up to 120 months
Comparison of PFS following initiation of larotrectinib to that following the line of therapy immediately preceding larotrectinib in each subject who has received prior therapy | Up to 120 months
Number of subjects with AEs categorized by severity. (including all, serious, and those considered treatment related.) | Up to 120 months
Number of subjects with safety-relevant changes in clinical parameters or vital signs after drug administration | Up to 120 months
Severity of safety-relevant changes in clinical parameters or vital signs after drug administration | Up to 120 months
Concordance coefficient | Up to 120 months
  Concordance of prior molecular profiling that detected an NTRK fusion within the subject's tumor with the diagnostic test being evaluated by the Sponsor.

CONTACTS AND LOCATIONS:
Locations (98):
- United States (18):
  - Stanford Cancer Center Palo Alto, Palo Alto, California
  - UCLA Health Santa Monica Cancer Care, Santa Monica, California
  - Memorial Cancer Institute at West, Pembroke Pines, Florida
  - The University of Chicago Medical Center - Hyde Park - Hematology & Oncology, Chicago, Illinois
  - Mass General Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute - Oncology Department, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center New York - Main Campus, New York, New York
  - UNC Hospitals - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Cleveland Clinic - Neurology, Cleveland, Ohio
  - Sidney Kimmel Cancer Center - Jefferson Health, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Avera Cancer Institute - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center - Texas Medical Center, Houston, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Fred Hutch Cancer Center - Sloan Clinic 1, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
- Argentina (5):
  - Hospital Alemán, Buenos Aires, Ciudad Auton. de Buenos Aires
  - Centro Estudios Médicos e Invest. Clínicas "Dr. N. Quirno", Buenos Aires, Ciudad Auton. de Buenos Aires
  - Fundación Cenit para la Investigación en Neurociencias, CABA, Ciudad Auton. de Buenos Aires
  - Centro Medico Austral, TBC, Ciudad Auton. de Buenos Aires
  - Centro Médico San Roque, San Miguel de Tucumán, Tucumán Province
- Australia (3):
  - Macquarie University Hospital, Sydney, New South Wales
  - Royal Darwin Hospital, Tiwi, Northern Territory
  - St John of God Healthcare, Subiaco, Western Australia
- Institut Jules Bordet/Jules Bordet Instituut, Brussels, Belgium
- Brazil (10):
  - Hosp. Araujo Jorge da Associação de Combate ao Câncer, Goiânia, Goiás
  - Cenantron Centro Avançado de Tratamento Oncológico, Ltda., Belo Horizonte, Minas Gerais
  - Fundacao Pio XII - Hospital de Cancer de Barretos, Barretos/SP, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo, São Paulo, São Paulo
  - Real e Benemérita Associação Portuguesa de Beneficência, São Paulo, São Paulo
  - IBCC - Instituto Brasileiro de Controle do Cancer, São Paulo, São Paulo
  - Instituto Nacional do Câncer - INCA - HC II, Rio de Janeiro
  - INCA - Hospital do Cancer III, Rio de Janeiro
  - Oncoclínicas Rio de Janeiro S.A, Rio de Janeiro
  - Hospital Sirio Libanes, São Paulo
- Tom Baker Cancer Centre, Calgary, Alberta, Canada
- China (4):
  - Beijing Cancer Hospital - Oncology Department, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Sichuan University West China Hospital, Chengdu, Sichuan
  - Zhongshan Hospital, Fudan University - Oncology Department, Shanghai
- Colombia (3):
  - Instituto Nacional de Cancerología INC Colombia, Bogota, Cundinamarca
  - Oncomédica S.A., Montería, Departamento de Córdoba
  - Fundación Oftalmológica de Santander Carlos Ardila Lule, Floridablanca, Santander Department
- Fakultní Nemocnice Olomouc, Olomouc, Czechia
- Rigshospitalet - Kræftbehandling, Copenhagen OE, Denmark
- France (8):
  - Hopital Jean Minjoz, Besançon
  - Institut Bergonie - Unicancer Nouvelle Aquitaine - Service Oncologie medicale, Bordeaux
  - Centre Antoine Lacassagne - Departement Oncologie, Nice
  - Hopital Saint Antoine APHP - Departement Oncologie, Paris
  - APHP-Hopital la Pitie Salpetriere-Departement oncologie, Paris
  - Hôpital de la Milétrie, Poitiers
  - Institut de Cancerologie Ouest - Saint-Herblain, Saint-Herblain
  - ICANS - Institut de Cancerologie de Strasbourg Europe - service oncologie medicale, Strasbourg
- Charité Comprehensive Cancer Center (CCCC), Berlin, Germany
- India (2):
  - All India Institute of Medical Sciences, Bhubaneswar, Odisha
  - Jawaharlal Institute Of Postgraduate Medical Education and R, Gorimedu, Puducherry
- St Vincents University Hospital, Dublin, Ireland
- Italy (6):
  - A.O.R.N. San Giuseppe Moscati, Avellino, Campania
  - A.O.U. di Bologna Policlinico S.Orsola Malpighi, Bologna, Emilia-Romagna
  - A.S.U. Friuli Centrale - A. Regionale Coordinamento Salute, Udine, Friuli Venezia Giulia
  - IRCCS Istituti Fisioterapici Ospitalieri - IFO, Rome, Lazio
  - Istituto Europeo di Oncologia s.r.l, Milan, Lombardy
  - Istituto Oncologico Veneto, Padua, Veneto
- Japan (4):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - The Cancer Institute Hospital of JFCR, Koto-ku, Tokyo
- IPO Porto, Porto, Portugal
- Russia (6):
  - Arkhangelsk Clinical Oncology Dispensary, Arkhangelsk
  - Republican Clinical Oncology Dispensary Kazan, Kazan'
  - Russian Oncological Scientific Center n.a. N.N. Blokhin RAMS, Moscow
  - 1st Moscow State Medical University n.a. I.M.Sechenov, Moscow
  - Clinical Diagnostical Center, Nizhny Novgorod
  - St. Petersburg Clinical Onc. Cent. of Spec. Types of Care, Saint Petersburg
- National Cancer Center Singapore - Oncology Department, Singapore, Singapore
- Slovakia (2):
  - Onkologicky Ustav Svatej Alzbety, s.r.o., Bratislava
  - Narodny onkologicky ustav, Bratislava
- South Korea (4):
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center-Ophthalmology, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center - Oncology Department, Seoul
- Spain (6):
  - Institut Catala D'oncologia - Oncologia, Barcelona, L Hospitalet de Llobregat
  - Hospital del Mar, Barcelona
  - Ciutat Sanitaria i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Maranon | Oncologia, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Centro Integral Oncológico Clara Campal, Madrid
- Karolinska Universitetssjukhuset Solna - Tema Cancer, Stockholm, Sweden
- Tri-Service General Hospital, Taipei, Taiwan
- Turkey (Türkiye) (7):
  - Health Ministry Of Türkiye Republic Ankara Bilkent City Hospital, Ankara
  - Trakya Univ. Tip Fak., Edirne
  - Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul
  - Istanbul Universitesi Cerrahpasa-Cerrahpasa Tip Fakultesi, Istanbul
  - TC Saglik Bakanligi Goztepe ProfDr Suleyman Yalcin Sehir Has, Istanbul
  - Izmir Katip Celebi Universitesi Ataturk Egitim ve Arastirma, Izmir
  - Erciyes Universitesi Tip Fakultesi, Kayseri

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Background] Waguespack SG, Drilon A, Lin JJ, Brose MS, McDermott R, Almubarak M, Bauman J, Casanova M, Krishnamurthy A, Kummar S, Leyvraz S, Oh DY, Park K, Sohal D, Sherman E, Norenberg R, Silvertown JD, Brega N, Hong DS, Cabanillas ME. Efficacy and safety of larotrectinib in patients with TRK fusion-positive thyroid carcinoma. Eur J Endocrinol. 2022 Apr 29;186(6):631-643. doi: 10.1530/EJE-21-1259. PMID 35333737
- [Derived] Brose MS, Westphalen CB, Pan X, Bernard-Gauthier V, Kurtinecz M, Guo H, Aris V, Brett NR, Majdi A, Subbiah V, Pennell NA, Kehl KL, Drilon A. Larotrectinib Compared With Real-World Non-Tropomyosin Receptor Kinase Inhibitor Therapies in Patients With Tropomyosin Receptor Kinase Fusion Cancer. JCO Precis Oncol. 2025 Apr;9:e2400500. doi: 10.1200/PO-24-00500. Epub 2025 Apr 23. PMID 40267388
- [Derived] Mascarenhas L, DuBois SG, Albert CM, Bielack S, Orbach D, Federman N, Geoerger B, Nagasubramanian R, Zhang Y, Chisholm J, Gallego Melcon S, Goto H, Morgenstern DA, Owens C, Pappo AS, Perreault S, Schulte JH, Shukla N, Zwaan CM, Neu N, Bernard-Gauthier V, De La Cuesta E, van Tilburg CM, Laetsch TW. Elective Discontinuation of Larotrectinib in Pediatric Patients With TRK Fusion Sarcomas and Related Mesenchymal Tumors. J Clin Oncol. 2025 Apr;43(10):1180-1187. doi: 10.1200/JCO.24.00848. Epub 2025 Jan 27. PMID 39869835
- [Derived] Hsieh CY, Hsu FL, Tsai TF. Comparison of Drug-Free Remission after the End of Phase III Trials of Three Different Anti-IL-23 Inhibitors in Psoriasis. Dermatol Ther (Heidelb). 2024 Sep;14(9):2607-2620. doi: 10.1007/s13555-024-01229-6. Epub 2024 Jul 29. PMID 39073712
- [Derived] Subbiah V, Burris HA 3rd, Kurzrock R. Revolutionizing cancer drug development: Harnessing the potential of basket trials. Cancer. 2024 Jan;130(2):186-200. doi: 10.1002/cncr.35085. Epub 2023 Nov 7. PMID 37934000
- [Derived] Kummar S, Shen L, Hong DS, McDermott R, Keedy VL, Casanova M, Demetri GD, Dowlati A, Melcon SG, Lassen UN, Leyvraz S, Liu T, Moreno V, Patel J, Patil T, Mallick AB, Sousa N, Tahara M, Ziegler DS, Norenberg R, Arvis P, Brega N, Drilon A, Tan DSW. Larotrectinib efficacy and safety in adult patients with tropomyosin receptor kinase fusion sarcomas. Cancer. 2023 Dec 1;129(23):3772-3782. doi: 10.1002/cncr.35036. Epub 2023 Sep 28. PMID 37769113
- [Derived] Bokemeyer C, Paracha N, Lassen U, Italiano A, Sullivan SD, Marian M, Brega N, Garcia-Foncillas J. Survival Outcomes of Patients With Tropomyosin Receptor Kinase Fusion-Positive Cancer Receiving Larotrectinib Versus Standard of Care: A Matching-Adjusted Indirect Comparison Using Real-World Data. JCO Precis Oncol. 2023 Jan;7:e2200436. doi: 10.1200/PO.22.00436. PMID 36689698
- [Derived] Rudzinski ER, Drilon A, Moore A, Spinosa S, Willi M, Laetsch TW. Testing methods to diagnose TRK fusion cancer - a plain language summary and patient perspective. Future Oncol. 2022 Dec;18(38):4141-4151. doi: 10.2217/fon-2022-0863. Epub 2023 Jan 6. PMID 36606522
- [Derived] Le X, Baik C, Bauman J, Gilbert J, Brose MS, Grilley-Olson JE, Patil T, McDermott R, Raez LE, Johnson JM, Shen L, Tahara M, Ho AL, Norenberg R, Dima L, Brega N, Drilon A, Hong DS. Larotrectinib Treatment for Patients With TRK Fusion-Positive Salivary Gland Cancers. Oncologist. 2022 May 10;29(6):e779-88. doi: 10.1093/oncolo/oyac080. Online ahead of print. PMID 35536733
- [Derived] Drilon A, Tan DSW, Lassen UN, Leyvraz S, Liu Y, Patel JD, Rosen L, Solomon B, Norenberg R, Dima L, Brega N, Shen L, Moreno V, Kummar S, Lin JJ. Efficacy and Safety of Larotrectinib in Patients With Tropomyosin Receptor Kinase Fusion-Positive Lung Cancers. JCO Precis Oncol. 2022 Jan;6:e2100418. doi: 10.1200/PO.21.00418. PMID 35085007
- [Derived] Doz F, van Tilburg CM, Geoerger B, Hojgaard M, Ora I, Boni V, Capra M, Chisholm J, Chung HC, DuBois SG, Gallego-Melcon S, Gerber NU, Goto H, Grilley-Olson JE, Hansford JR, Hong DS, Italiano A, Kang HJ, Nysom K, Thorwarth A, Stefanowicz J, Tahara M, Ziegler DS, Gavrilovic IT, Norenberg R, Dima L, De La Cuesta E, Laetsch TW, Drilon A, Perreault S. Efficacy and safety of larotrectinib in TRK fusion-positive primary central nervous system tumors. Neuro Oncol. 2022 Jun 1;24(6):997-1007. doi: 10.1093/neuonc/noab274. PMID 34850167
- [Derived] Lee YA, Lee H, Im SW, Song YS, Oh DY, Kang HJ, Won JK, Jung KC, Kwon D, Chung EJ, Hah JH, Paeng JC, Kim JH, Choi J, Kim OH, Oh JM, Ahn BC, Wirth LJ, Shin CH, Kim JI, Park YJ. NTRK and RET fusion-directed therapy in pediatric thyroid cancer yields a tumor response and radioiodine uptake. J Clin Invest. 2021 Sep 15;131(18):e144847. doi: 10.1172/JCI144847. PMID 34237031
- [Derived] Bebb DG, Banerji S, Blais N, Desmeules P, Gill S, Grin A, Feilotter H, Hansen AR, Hyrcza M, Krzyzanowska M, Melosky B, Noujaim J, Purgina B, Ruether D, Simmons CE, Soulieres D, Torlakovic EE, Tsao MS. Canadian Consensus for Biomarker Testing and Treatment of TRK Fusion Cancer in Adults. Curr Oncol. 2021 Jan 15;28(1):523-548. doi: 10.3390/curroncol28010053. PMID 33467570
- [Derived] Perreault S, Chami R, Deyell RJ, El Demellawy D, Ellezam B, Jabado N, Morgenstern DA, Narendran A, Sorensen PHB, Wasserman JD, Yip S. Canadian Consensus for Biomarker Testing and Treatment of TRK Fusion Cancer in Pediatric Patients. Curr Oncol. 2021 Jan 9;28(1):346-366. doi: 10.3390/curroncol28010038. PMID 33435412
- [Derived] Hong DS, DuBois SG, Kummar S, Farago AF, Albert CM, Rohrberg KS, van Tilburg CM, Nagasubramanian R, Berlin JD, Federman N, Mascarenhas L, Geoerger B, Dowlati A, Pappo AS, Bielack S, Doz F, McDermott R, Patel JD, Schilder RJ, Tahara M, Pfister SM, Witt O, Ladanyi M, Rudzinski ER, Nanda S, Childs BH, Laetsch TW, Hyman DM, Drilon A. Larotrectinib in patients with TRK fusion-positive solid tumours: a pooled analysis of three phase 1/2 clinical trials. Lancet Oncol. 2020 Apr;21(4):531-540. doi: 10.1016/S1470-2045(19)30856-3. Epub 2020 Feb 24. PMID 32105622
- [Derived] O'Reilly EM, Hechtman JF. Tumour response to TRK inhibition in a patient with pancreatic adenocarcinoma harbouring an NTRK gene fusion. Ann Oncol. 2019 Nov 1;30(Suppl_8):viii36-viii40. doi: 10.1093/annonc/mdz385. Epub 2019 Dec 24. PMID 31605106
- [Derived] Drilon A, Laetsch TW, Kummar S, DuBois SG, Lassen UN, Demetri GD, Nathenson M, Doebele RC, Farago AF, Pappo AS, Turpin B, Dowlati A, Brose MS, Mascarenhas L, Federman N, Berlin J, El-Deiry WS, Baik C, Deeken J, Boni V, Nagasubramanian R, Taylor M, Rudzinski ER, Meric-Bernstam F, Sohal DPS, Ma PC, Raez LE, Hechtman JF, Benayed R, Ladanyi M, Tuch BB, Ebata K, Cruickshank S, Ku NC, Cox MC, Hawkins DS, Hong DS, Hyman DM. Efficacy of Larotrectinib in TRK Fusion-Positive Cancers in Adults and Children. N Engl J Med. 2018 Feb 22;378(8):731-739. doi: 10.1056/NEJMoa1714448. PMID 29466156
- [Derived] Shi E, Chmielecki J, Tang CM, Wang K, Heinrich MC, Kang G, Corless CL, Hong D, Fero KE, Murphy JD, Fanta PT, Ali SM, De Siena M, Burgoyne AM, Movva S, Madlensky L, Heestand GM, Trent JC, Kurzrock R, Morosini D, Ross JS, Harismendy O, Sicklick JK. FGFR1 and NTRK3 actionable alterations in "Wild-Type" gastrointestinal stromal tumors. J Transl Med. 2016 Dec 14;14(1):339. doi: 10.1186/s12967-016-1075-6. PMID 27974047